CLINICAL TRIAL: NCT03088956
Title: A Study to Model Rates of Change on Neuropsychological Test Measures in Subjects Diagnosed With Behavioral Variant Frontotemporal Dementia and Healthy Subjects
Brief Title: Cognitive, Behavioral, and Functional Change in Behavioral Variant Frontotemporal Dementia (bvFTD)
Acronym: FORWARD
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 992FD001
Record Dates: First submitted 2017-03-17; First posted 2017-03-24 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Frontotemporal Dementia; Behavioral Variant Frontotemporal Dementia
Keywords: Longitudinal; Caregiver; Cognitive assessments; Behavioral assessments; Functional assessments
MeSH Terms: conditions — Frontotemporal Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- bvFTD: Participants with behavioral variant frontotemporal dementia (bvFTD) (n=37)
  Interventions: Other: Assessments
- Healthy: Healthy Participants (n=10)
  Interventions: Other: Assessments

INTERVENTIONS:
Other: Assessments — Cognitive, Behavioral and Functional as described in the Outcome Measures

SUMMARY:
The objectives of the study are to; (1) estimate the change in disease -related cognitive decline over 1 year on a battery of cognitive tests administered to participants with early-stage symptomatic Behavioral Variant Frontotemporal Dementia (bvFTD) phenotypic variant; (2) identify the cognitive test or brief battery of cognitive tests which are the most sensitive to detect bvFTD progression; (3) determine the optimal schedule of administration of cognitive tests to detect bvFTD progression; (4) evaluate the relationship between cognitive tests and measures of behavior, function, caregiver's burden, quality of life (QOL); and (5) obtain blood samples for genetic and exploratory biomarkers correlations.

ELIGIBILITY:
Key Inclusion Criteria for Participants with behavioral variant frontotemporal dementia (bvFTD):

* Must speak and understand oral and written English.
* Must have probable bvFTD.
* Must have a global Clinical Dementia Rating (CDR) score of 0.5-1 and a Mini Mental State Examination (MMSE) score ≥20 to reflect early stages of disease.
* Must have 1 informant/caregiver who, in the Investigator's judgment, has frequent and sufficient contact with the participant as to be able to provide accurate information about the participant's behaviors as well as cognitive and functional abilities.
* Must be ambulatory or able to walk with assistance and not be institutionalized.

Key Inclusion Criteria for Healthy Participants:

* Must speak and understand oral and written English.
* Must be in good general health determined by Investigator.

Key Exclusion Criteria for Participants with bvFTD:

* Concomitant motor neuron disease with limb or bulbar weakness which, in the opinion of the Investigator, may affect performance over the course of the study. Participants with bvFTD with motor neuron disease are otherwise allowed to participate.
* Known presence of a structural brain lesion that could reasonably explain symptoms.
* Diagnosis of Alzheimer's disease and/or known presence of an Alzheimer's disease causing mutation in PSEN1, PSEN2 or APP; or neuropathological evidence for Alzheimer's disease as a cause of syndrome.
* History of other acute or chronic neurological or psychiatric conditions that are unrelated and may confound a diagnosis of bvFTD and that, in the opinion of the Investigator, may affect cognition, behavior, or ability to complete the study.
* History of severe alcohol or substance abuse.
* History of disorders that could confound a diagnosis of bvFTD.
* Use of allowed chronic medications at doses that have not been stable for at least 4 weeks prior to Screening.
* Current use of psychoactive medication that will interfere with accurate assessment of cognition (as assessed by the Investigator)

Key Exclusion Criteria for Healthy Participants:

* History of alcohol or substance abuse.
* Current use of psychoactive medication that will interfere with accurate assessment of cognition (as assessed by the Investigator).

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Academic centers, Hospitals, Clinics
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Annualized rate of change in International Shopping List Test (ISLT) - Immediate Recall | Up to 12 Months
  ISLT uses a word list learning paradigm to measure verbal learning. The score for this test is based on the total number of correct responses made in remembering the list on 3 consecutive trials at a single session. Higher scores indicate better performance.
Annualized rate of change in Detection Test | Up to 12 Months
  A test that uses a simple reaction time paradigm to measure psychomotor function. The score for this test is based on the speed of performance, measured as the mean of the log10 transformed reaction times for correct responses. Lower scores indicate better performance.
Annualized rate of change in Identification Test | Up to 12 Months
  A test that uses a choice reaction time paradigm to measure attention. The score for this test is based on the speed of performance, measured as the mean of the log10 transformed reaction times for correct responses. Lower scores indicate better performance.
Annualized rate of change in One Back Test | Up to 12 Months
  A test that uses an n-back paradigm to measure working memory. The score for this test is based on the speed of performance, measured as the mean of the log10 transformed reaction times for correct responses. Lower scores indicate better performance.
Annualized rate of change in Groton Maze Learning Test | Up to 12 Months
  Modified version (10 x 10, "snake maze" version): this is a test that uses a maze learning paradigm to measure executive function and spatial learning. The score for this test is based on the total number of errors made in attempting to learn the same hidden pathway on 5 consecutive trials at a single session. Lower scores indicate better performance.
Annualized rate of change in ISLT - Delayed Recall | Up to 12 Months
  A test that uses a word list paradigm to measure verbal memory. The score for this test is based on the total number of correct responses made in remembering the list after a delay. Higher scores indicate better performance.
Annualized rate of change in Social Emotional Cognition Test (SECT) | Up to 12 Months
  A test that uses an odd-man-out paradigm to measure social cognition. The score for this test is based on the accuracy of performance, measured as the arcsine transformation of the square root of the proportion of correct responses. Higher scores indicate better performance.
Annualized rate of change in Letter Fluency | Up to 12 Months
  A test that assesses executive function by asking the participant to state as many words as possible starting with a specific letter. The score for this test is based on the number of words generated. Higher scores indicate better performance.
Annualized rate of change in Category Fluency | Up to 12 Months
  A test that assesses executive function by asking the participant to state as many words as possible within a given category. The score for this test is based on the number of words generated. Higher scores indicate better performance.
Annualized rate of change in Digit Symbol Coding (DSC) | Up to 12 Months
  A paper and pencil test that assesses attention, working memory, and executive function. The participant is presented with a paper on top of which is printed a key showing numerals paired with symbols and on the bottom are rows of numerals with a blank space beneath each one. The participant is instructed to draw the symbol that matches each numeral and to complete as many as possible in order in 2 minutes. The score for this test is the number of correct responses. Higher scores indicate better performance.
Annualized rate of change in Letter Number Sequencing (LNS) | Up to 12 Months
  A test that assesses working memory by asking the participant to recall series of numbers and letters presented in random order, but to respond by reciting the numbers in ascending order followed by letters in alphabetical order. The score for this test is based on the number of correct answers. Higher scores indicate better performance.
Annualized rate of change in Mini Mental State Examination (MMSE) | Up to 12 Months
  A test that assesses working memory by asking the participant to recall series of numbers and letters presented in random order, but to respond by reciting the numbers in ascending order followed by letters in alphabetical order. The score for this test is based on the number of correct answers. Higher scores indicate better performance.
Change from Day 1 in International Shopping List Test (ISLT) - Immediate Recall | Up to 12 Months
  ISLT uses a word list learning paradigm to measure verbal learning. The score for this test is based on the total number of correct responses made in remembering the list on 3 consecutive trials at a single session. Higher scores indicate better performance.
Change from Day 1 in Detection Test | Up to 12 Months
  A test that uses a simple reaction time paradigm to measure psychomotor function. The score for this test is based on the speed of performance, measured as the mean of the log10 transformed reaction times for correct responses. Lower scores indicate better performance.
Change from Day 1 in Identification Test | Up to 12 Months
  A test that uses a choice reaction time paradigm to measure attention. The score for this test is based on the speed of performance, measured as the mean of the log10 transformed reaction times for correct responses. Lower scores indicate better performance.
Change from Day 1 in One Back Test | Up to 12 Months
  A test that uses an n-back paradigm to measure working memory. The score for this test is based on the speed of performance, measured as the mean of the log10 transformed reaction times for correct responses. Lower scores indicate better performance.
Change from Day 1 in Groton Maze Learning Test | Up to 12 Months
  Modified version (10 x 10, "snake maze" version): this is a test that uses a maze learning paradigm to measure executive function and spatial learning. The score for this test is based on the total number of errors made in attempting to learn the same hidden pathway on 5 consecutive trials at a single session. Lower scores indicate better performance.
Change from Day 1 in ISLT- Delayed Recall | Up to 12 Months
  A test that uses a word list paradigm to measure verbal memory. The score for this test is based on the total number of correct responses made in remembering the list after a delay. Higher scores indicate better performance.
Change from Day 1 in SECT | Up to 12 Months
  A test that uses an odd-man-out paradigm to measure social cognition. The score for this test is based on the accuracy of performance, measured as the arcsine transformation of the square root of the proportion of correct responses. Higher scores indicate better performance.
Change from Day 1 in Letter Fluency | Up to 12 Months
  A test that assesses executive function by asking the participant to state as many words as possible starting with a specific letter. The score for this test is based on the number of words generated. Higher scores indicate better performance.
Change from Day 1 in Category Fluency | Up to 12 Months
  A test that assesses executive function by asking the participant to state as many words as possible within a given category. The score for this test is based on the number of words generated. Higher scores indicate better performance.
Change from Day 1 in DSC | Up to 12 Months
  A paper and pencil test that assesses attention, working memory, and executive function. The participant is presented with a paper on top of which is printed a key showing numerals paired with symbols and on the bottom are rows of numerals with a blank space beneath each one. The participant is instructed to draw the symbol that matches each numeral and to complete as many as possible in order in 2 minutes. The score for this test is the number of correct responses. Higher scores indicate better performance.
Change from Day 1 in LNS | Up to 12 Months
  A test that assesses working memory by asking the participant to recall series of numbers and letters presented in random order, but to respond by reciting the numbers in ascending order followed by letters in alphabetical order. The score for this test is based on the number of correct answers. Higher scores indicate better performance.
Change from Day 1 in MMSE | Up to 12 months
  A test that assesses working memory by asking the participant to recall series of numbers and letters presented in random order, but to respond by reciting the numbers in ascending order followed by letters in alphabetical order. The score for this test is based on the number of correct answers. Higher scores indicate better performance.
Actual values from Day 1 in Neurophsychic Inventory (NPI) | Up to 12 Months
  A 12-item participant and caregiver interview based questionnaire assessing behavioral domains which are common in dementia: hallucinations, delusions, agitation/aggression, dysphoria/depression, anxiety, irritability, disinhibition, euphoria, apathy, aberrant motor behavior, sleep and night-time behavior disorders, and appetite and eating disorders. Each domain is scored for frequency on a 4-item scale (1 = rarely to 4 = very often), for severity on a 3-item scale (1 = mild to 3 = severe), and for associated caregiver distress on a 6-item scale (0 = not at all to 5 = very severe or extremely).
Change from Day 1 in NPI | Up to 12 Months
  A 12-item participant and caregiver interview based questionnaire assessing behavioral domains which are common in dementia: hallucinations, delusions, agitation/aggression, dysphoria/depression, anxiety, irritability, disinhibition, euphoria, apathy, aberrant motor behavior, sleep and night-time behavior disorders, and appetite and eating disorders. Each domain is scored for frequency on a 4-item scale (1 = rarely to 4 = very often), for severity on a 3-item scale (1 = mild to 3 = severe), and for associated caregiver distress on a 6-item scale (0 = not at all to 5 = very severe or extremely).
Actual values from Day 1 in Neurophsychic Inventory Questionnaire (NPI-Q) | Up to 12 Months
  A shorter version of the NPI, intended for use in routine clinical practice. The NPI-Q contains 12 questions scored on symptom presence (yes/no) and severity (mild, moderate, and severe). Frequency on a 4-item scale (rarely to very often) and associated caregiver distress on a 6-item scale (0 = not at all to 5 = very severe or extreme) will also be collected.
Change from Day 1 in NPI-Q | Up to 12 Months
  A shorter version of the NPI, intended for use in routine clinical practice. The NPI-Q contains 12 questions scored on symptom presence (yes/no) and severity (mild, moderate, and severe). Frequency on a 4-item scale (rarely to very often) and associated caregiver distress on a 6-item scale (0 = not at all to 5 = very severe or extreme) will also be collected.
Actual values from Day 1 in Revised Self-Monitoring Scale | Up to 12 Months
  A 13-item version of the Self-Monitoring Scale [Snyder 1974] which measures sensitivity to the expressive behavior of others and ability to modify self-presentation.
Change from Day 1 in Revised Self-Monitoring Scale | Up to 12 Months
  A 13-item version of the Self-Monitoring Scale [Snyder 1974] which measures sensitivity to the expressive behavior of others and ability to modify self-presentation.
Actual values from Day 1 in Apathy Inventory | Up to 12 Months
  Assesses 3 dimensions of apathy: emotional blunting, lack of initiative, and lack of interest, with 1 version each for participants, caregivers, and clinicians. Higher scores reflect greater apathy. For the participant version, yes/no responses are captured for each dimension, then a visual analogue scale or numeric evaluation from 1-12 is captured for severity of functioning (1=mild to 12=extremely severe), for a total score of 36. For the caregiver version, each dimension is scored on a 12-point Likert scale based on frequency (1=occasionally to 4=very frequently: and severity (1=mild to 3=marked), for a total score of 36. The clinician version captures each domain on a scale from 0 to 4 (0=no problem to 4=major problem), for a total score of 12.
Change from Day 1 in Apathy Inventory | Up to 12 Months
  Assesses 3 dimensions of apathy: emotional blunting, lack of initiative , and lack of interest , with 1 version each for participants, caregivers, and clinicians. Higher scores reflect greater apathy. For the participant version, yes/no responses are captured for each dimension, then a visual analogue scale or numeric evaluation from 1-12 is captured for severity of functioning (1=mild to 12=extremely severe), for a total score of 36. For the caregiver version, each dimension is scored on a 12-point Likert scale based on frequency (1=occasionally to 4=very frequently: and severity (1=mild to 3=marked), for a total score of 36. The clinician version captures each domain on a scale from 0 to 4 (0=no problem to 4=major problem), for a total score of 12.
Actual values from Day 1 in Family Accommodation Scale for Obsessive Compulsive Disorder - Self Rated (FAS-SR) | Up to 12 Months
  This is a self-rated version of the Family Accommodation Scale for Obsessive Compulsive Disorder to be completed by the caregiver, which assesses the number of days with accommodating behaviors in the past week using a 5-point Likert scale (0 = none to 4 = every day).
Change from Day 1 in FAS-SR | Up to 12 Months
  This is a self-rated version of the Family Accommodation Scale for Obsessive Compulsive Disorder to be completed by the caregiver, which assesses the number of days with accommodating behaviors in the past week using a 5-point Likert scale (0 = none to 4 = every day).
Actual values from Day 1 in Behavior Rating Scale | Up to 12 Months
  A questionnaire completed by the clinic rater assessing participant's behaviors on a 4-item severity scale (none to severe). Behaviors include agitation, stimulus boundedness, perseverative behavior, decreased initiation, motor stereotypies, distractibility, lack of social/emotional engagement, impulsivity, socially inappropriateness, and impaired or fluctuating levels of alertness.
Change from Day 1 in Behavior Rating Scale | Up to 12 Months
  A questionnaire completed by the clinic rater assessing participant's behaviors on a 4-item severity scale (none to severe). Behaviors include agitation, stimulus boundedness, perseverative behavior, decreased initiation, motor stereotypies, distractibility, lack of social/emotional engagement, impulsivity, socially inappropriateness, and impaired or fluctuating levels of alertness.
Actual values from Day 1 in Functional Activities Questionnaire (FAQ) | Up to 12 Months
  A 10-item questionnaire designed to assess independence in participants with Alzheimer's Disease by measuring instrumental activities of daily living. Each question is rated on a 4-point Likert scale (0 = normal to 3 = dependent).
Change from Day 1 in FAQ | Up to 12 Months
  A 10-item questionnaire designed to assess independence in participants with Alzheimer's Disease by measuring instrumental activities of daily living. Each question is rated on a 4-point Likert scale (0 = normal to 3 = dependent).
Actual values from Day 1 in Clinical Global Impression of Change (CGIC) | Up to 12 Months
  This is 1 of the items of the Clinical Global Impression, and measures clinical change as improvement or worsening. It is scored on a 7-point Likert scale (marked improvement to no change and to marked worsening).
Change from Day 1 in CGIC | Up to 12 Months
  This is 1 of the items of the Clinical Global Impression, and measures clinical change as improvement or worsening. It is scored on a 7-point Likert scale (marked improvement to no change and to marked worsening).
Actual values from Day 1 in Clinical Dementia Rating-Frontotemporal Lobar Degeneration (CDR-FTLD) | Up to 12 Months
  An FTLD-modified CDR scale (initially developed for Alzheimer's Disease) which includes 2 additional domains: behavior/comportment/personality and language, to the CDR 6 domains: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. Each domain is scored on a 5-point impairment Likert scale (normal to severe dementia).
Change from Day 1 in CDR-FTLD | Up to 12 Months
  An FTLD-modified CDR scale (initially developed for Alzheimer's Disease) which includes 2 additional domains: behavior/comportment/personality and language, to the CDR 6 domains: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. Each domain is scored on a 5-point impairment Likert scale (normal to severe dementia).
Actual values from Day 1 in Unified Parkinson's Disease Rating Scale (UPDRS) Part III | Up to 12 Months
  A motor examination domain of the UPDRS, designed to assess progression of Parkinson's disease. It consists of 14 questions scored on a 5-point severity Likert scale (0 to 4).
Change from Day 1 in UPDRS Part III | Up to 12 Months
  A motor examination domain of the UPDRS, designed to assess progression of Parkinson's disease. It consists of 14 questions scored on a 5-point severity Likert scale (0 to 4).
Actual values from Day 1 of caregiver's Quality of Life (QOL) in Zarit Caregiver Burden Interview | Up to 12 Months
  A caregiver self-reported measure to assess level of burden when taking care of someone, consisting of a 22-item questionnaire. Each question is scored on a 5-point Likert scale (0 = never to 4 = nearly always).
Change from Day 1 of caregiver's QOL in Zarit Caregiver Burden Interview | Up to 12 Months
  A caregiver self-reported measure to assess level of burden when taking care of someone, consisting of a 22-item questionnaire. Each question is scored on a 5-point Likert scale (0 = never to 4 = nearly always).
Actual values from Day 1 of QOL in Geriatric Depression Scale- Short Form (GDS-SF) | Up to 12 Months
  A 15-item questionnaire developed to assess depression symptoms in elderly participants (55 years or older). Each question is scored as yes/no. This measure has been used in similar dementia populations, such as Alzheimer's and Parkinson's, in addition to 1 FTD study [Matsuzono 2015]. While the population in this study may be a bit younger, this measure will be tested for use in the bvFTD population included.
Change from Day 1 of QOL in GDS-SF | Up to 12 Months
  A 15-item questionnaire developed to assess depression symptoms in elderly participants (55 years or older). Each question is scored as yes/no. This measure has been used in similar dementia populations, such as Alzheimer's and Parkinson's, in addition to 1 FTD study [Matsuzono 2015]. While the population in this study may be a bit younger, this measure will be tested for use in the bvFTD population included.
Actual values from Day 1 of caregiver's QOL in Caregiver Assessment Measure | Up to 12 Months
  A questionnaire developed by Biogen which consists of 4 questions. The first 2 questions are scored on a 5-point Likert scale (0 = not at all to 4 = a great deal) and refer to the impact of the participant's disease on the caregiver. The third question refers to the change in the participant's need of care; in case this has increased, an additional question is to be scored on a 5-point Likert scale (0 = a little more care to 4 = a great deal more care). The last question refers to the amount of care (hours per day).
Change from Day 1 of caregiver's QOL in Caregiver Assessment Measure | Up to 12 Months
  A questionnaire developed by Biogen which consists of 4 questions. The first 2 questions are scored on a 5-point Likert scale (0 = not at all to 4 = a great deal) and refer to the impact of the participant's disease on the caregiver. The third question refers to the change in the participant's need of care; in case this has increased, an additional question is to be scored on a 5-point Likert scale (0 = a little more care to 4 = a great deal more care). The last question refers to the amount of care (hours per day).
Actual values from Day 1 of QOL in Quality of Life in Neurological Disorders (NeuroQOL) | Up to 12 Months
  A self-reported health-related quality of life (HRQL) assessment for adults with a neurological disorder, which measures 3 areas: physical health, mental health, and social health. All NeuroQOL items have 5 response options (1 = not at all to 5 = very much). Higher scores represent more impairment or worse health. Participants with bvFTD will complete the following sections of the NeuroQOL: Cognitive Function SF, Emotional and Behavioral Dyscontrol SF and Ability to Participate in Social Roles and Activities SF. Caregivers will complete the following sections of the NeuroQOL: Satisfaction with Social Roles SF and Activities and Ability to Participate in Social Roles and Activities SF.
Change from Day 1 of QOL in Quality of Life in NeuroQOL | Up to 12 Months
  A self-reported health-related quality of life (HRQL) assessment for adults with a neurological disorder, which measures 3 areas: physical health, mental health, and social health. All NeuroQOL items have 5 response options (1 = not at all to 5 = very much). Higher scores represent more impairment or worse health. Participants with bvFTD will complete the following sections of the NeuroQOL: Cognitive Function SF, Emotional and Behavioral Dyscontrol SF and Ability to Participate in Social Roles and Activities SF. Caregivers will complete the following sections of the NeuroQOL: Satisfaction with Social Roles SF and Activities and Ability to Participate in Social Roles and Activities SF.
Actual values from Day 1 of QOL in EuroOol 5 Dimensions Questionnaire (EQ-5D) | Up to 12 Months
  A self-reported generic HRQL assessment with 2 parts, the first containing 5 tick boxes (no problems, some problems, moderate problems, severe problems, cannot do) to select the most appropriate statement on each of its 5 domains (mobility, self care, usual activities, anxiety/ depression, and pain), and the second with a visual analogue scale ranging from "the best health you can imagine" to "the worst health you can imagine". This version with 5 response levels is called the EQ-5D-5L.
Change from Day 1 of QOL in EQ-5D | Up to 12 Months
  A self-reported generic HRQL assessment with 2 parts, the first containing 5 tick boxes (no problems, some problems, moderate problems, severe problems, cannot do) to select the most appropriate statement on each of its 5 domains (mobility, self care, usual activities, anxiety/ depression, and pain), and the second with a visual analogue scale ranging from "the best health you can imagine" to "the worst health you can imagine". This version with 5 response levels is called the EQ-5D-5L.
Actual values from Day 1 of QOL in Affect and Activity Indicators of QOL (AAIQOL) | Up to 12 Months
  A measure of caregiver-reported (proxy) QOL in participants with dementia which assesses 2 domains: activity and affect. Activity is a 15-item questionnaire rated on opportunity (no/yes), frequency (none/few/often), and enjoyment (yes/no), with 5 items for outdoors activities and 10 items for home activities. Affect is a 6-item questionnaire, with 3 items for positive effects and 3 items for negative effects, referring to the previous 2 weeks, and scored on a 5-point Likert scale (1 = never to 5 = several [3+] times per day).
Change from Day 1 of QOL in AAIQOL | Up to 12 Months
  A measure of caregiver-reported (proxy) QOL in participants with dementia which assesses 2 domains: activity and affect. Activity is a 15-item questionnaire rated on opportunity (no/yes), frequency (none/few/often), and enjoyment (yes/no), with 5 items for outdoors activities and 10 items for home activities. Affect is a 6-item questionnaire, with 3 items for positive effects and 3 items for negative effects, referring to the previous 2 weeks, and scored on a 5-point Likert scale (1 = never to 5 = several [3+] times per day).
Actual values from Day 1 for exploratory biomarkers | Baseline, Month 12
  Venipuncture for collection of whole blood samples for exploratory blood biomarkers analyses.
Change from Day 1 for exploratory blood biomarkers | Baseline, Month 12
  Venipuncture for collection of whole blood samples for exploratory blood biomarkers analyses.
bvFTD genetic mutations identification in whole blood samples | Baseline, Month 12
  Venipuncture for collection of whole blood samples for identification of bvFTD genetic mutations.
Potential identification of genetic biomarkers associated with bvFTD from DNA/RNA in whole blood samples | Baseline, Month 12
  Venipuncture for collection of whole blood samples for potential identification of genetic biomarkers associated with bvFTD.
Actual values at Day 1 in Clinical Global Impression of Severity (CGIS) | Day 1
  This is one of the items of the Clinical Global Impression, and measures clinical severity at baseline. It is rated on a 7-point Likert scale, with illness being rated in the range of 1 (normal) to 7 (severely ill). It requires the clinician to rate the severity of the participant's illness at the time of the assessment, relative to the clinician's past experience with participants who have the same diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (11):
- United States (11):
  - Research Site, Birmingham, Alabama
  - Research Site, Los Angeles, California
  - Research Site, Boca Raton, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Elk Grove Village, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Rochester, Minnesota
  - Research Site, Columbus, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Knoxville, Tennessee
  - Research Site, Seattle, Washington